CLINICAL TRIAL: NCT02254616
Title: Hybrid Approach to Mirror Therapy and Transcranial Direct Current Stimulation for Stroke Recovery: A Follow up Study on Brain Reorganization, Motor Performance of Upper Extremity, Daily Function, and Activity Participation
Brief Title: Hybrid Approach to Mirror Therapy and Transcranial Direct Current Stimulation for Stroke Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102-5696A3
Record Dates: First submitted 2014-09-16; First posted 2014-10-02 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke Rehabilitation; Hybrid therapy; Mirror Therapy; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mirror therapy with tDCS (Experimental): Functional training will consist of unilateral and bilateral functional tasks in daily living, and last for 30 minutes. Some examples are mopping the table by using the affected hand or scooping beans from a bowl with one hand while the other hand stabilizes the bowl. The principles of part-task practice and whole-task practice will be applied based on the participant's performance level.Functional training will consist of unilateral and bilateral functional tasks in daily living, and last for 30 minutes. Some examples are mopping the table by using the affected hand or scooping beans from a bowl with one hand while the other hand stabilizes the bowl. The principles of part-task practice and whole-task practice will be applied based on the participant's performance level.
  Interventions: Behavioral: Mirror Therapy with tDCS
- Mirror Therapy (Active Comparator): The MT only group will receive a 60-minute MT per session followed by a 30-minute functional training. Participant will go through the same protocol as that for the MT+tDCS and MT+sham tDCS groups with no tDCS presented in setting. This group is for evaluating placebo effect of the present of tDCS application.
  Interventions: Behavioral: Mirror Therapy
- Control Intervention (Active Comparator): The CI group will receive a 60-minute conventional stroke rehabilitation training followed by a 30-minute functional training. During the 60-mimute conventional training, interventions will include passive range of movement and muscle tone normalization techniques of the affected arm, and gross motor training (e.g., shoulder ladder activity), fine motor training (e.g., grasping cones), and muscle strength training in a unilateral and bilateral manners. During the 30-minute functional training, the same principles to those in the MT groups will be applied.
  Interventions: Behavioral: Control Intervention
- Mirror Therapy with sham-tDCS (Active Comparator): Functional training will consist of unilateral and bilateral functional tasks in daily living, and last for 30 minutes. Some examples are mopping the table by using the affected hand or scooping beans from a bowl with one hand while the other hand stabilizes the bowl. The principles of part-task practice and whole-task practice will be applied based on the participant's performance level.
  Interventions: Behavioral: Mirror Therapy with sham-tDCS

INTERVENTIONS:
Behavioral: Mirror Therapy with tDCS — The MTtDCS group will receive a 20-minute tDCS at 1.5 mA current intensity per session followed by a 40-minute mirror therapy and 30-minute functional training during the first two weeks. Sixty-minute pure mirror therapy during the last 2 weeks, and followed by a 30-minute functional training.
  Other Names: MTtDCS
  Arms: Mirror therapy with tDCS
Behavioral: Mirror Therapy with sham-tDCS — The MTtDCS(m) group will receive a 20-minute sham-tDCS per session followed by a 40-minute mirror therapy and 30-minute functional training during the first two weeks. Sixty-minute pure mirror therapy during the last 2 weeks, and followed by a 30-minute functional training.
  Other Names: MTtDCS(m)
  Arms: Mirror Therapy with sham-tDCS
Behavioral: Mirror Therapy — The MT group will receive a 60-minute MT per session followed by a 30-minute functional training.
  Other Names: MT
  Arms: Mirror Therapy
Behavioral: Control Intervention — The CI group will receive a 60-minute conventional stroke rehabilitation training followed by a 30-minute functional training.
  Other Names: CI
  Arms: Control Intervention

SUMMARY:
We hypothesize that (1) the hybrid therapy will induce greater improvements on some health-related outcomes compared to other therapies; (2) such benefits will retain at 6-month follow-up; (3) better motor control and brain reorganization will be found in the hybrid therapy than the other therapies; (4) correlations will be found between brain activity and movement kinematics/health-related outcomes.

DETAILED DESCRIPTION:
Chronic stroke participants will be recruited from the Chang Gung Memorial Hospital and then were randomly assigned to 1 of the 4 groups: MT+tDCS, MT+sham tDCS, MT, and CI groups. The participants in each group receive equivalent amounts of treatment.

Analysis of covariance (ANCOVA), controlling for the pretest differences, will be separately performed for each outcome measure to test the effects of different intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* First episode of stroke in cortical regions
* Time since stroke more than 6 months
* Initial motor part of UE of FMA score ranging from 24 to 52, indicating moderate to mild movement impairment
* No severe spasticity in any joints of the affected arm (Modified Ashworth Scale ≤ 2)
* No serious cognitive impairment (i.e., Mini Mental State Exam score≧ 24)
* Willing to sign the informed consent form.

Exclusion Criteria:

* Aphasia that might interfere with understanding instructions
* Visual/attention impairments that might interfere with the seeing of mirror illusion, including hemineglect/hemianopsia
* Major health problems or poor physical conditions that might limit participation
* Currently participation in any other research
* Previous brain neurosurgery
* Metallic implants within the brain.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Change scores of Fugl-Meyer Assessment (FMA) | Baseline, 2 weeks, 4 weeks, 16 weeks, and 28 weeks
  The upper-extremity subscale of the FMA will be used to assess motor impairment. The 33 upper limb items measure the movement and reflexes of the shoulder/elbow/forearm, wrist, hand, and coordination/speed. They are scored on a 3-point ordinal scale (0-cannot perform, 1-performs partially, 2-performs fully). The maximum score is 66, indicating optimal recovery. The sub-score of a proximal shoulder/elbow (FMA s/e: 0-42) and a distal hand/wrist (FMA h/w: 0-24) will be also calculated to investigate the treatment effects on separate upper extremity elements. The reliability, validity, and responsiveness of the FMA in stroke patients have been shown to be good.
Change scores of Wolf Motor Function Test (WMFT) | Baseline, 2 weeks, and 4 weeks
  The assessment requires the participant to perform 15 function-based and 2 strength-based tasks. The tasks are averaged to produce a score in seconds that ranges from 0 to 120 seconds. For functional ability scoring, we used a 6-point ordinal scale where 0 indicates "does not attempt with the involved arm" and 5 indicates "arm does participate; movement appears to be normal." The clinimetrics of the WMFT has been ascertained in stroke patients (Wolf et al., 2005).
Change scores of Motor Activity Log (MAL) | Baseline, 2 weeks, and 4 weeks, 16 weeks, and 28 weeks
  The MAL consists of 30 structured questions to interview how the patients rate the frequency (amount of use subscale) and quality (quality of movement subscale) of movements while using their affected arm to accomplish each of the 30 daily activities. The score of each item ranges from 0 to 5, and the higher scores indicate more frequently used or higher quality of movements. The clinimetric properties of the MAL in stroke patients have been validated (Uswatte, Taub, Morris, Light, & Thompson, 2006).
Change scores of Stroke Impact Scale Version 3.0 (SIS 3.0) | Baseline, 2 weeks, and 4 weeks, 16 weeks, and 28 weeks
  The SIS 3.0 is a stroke-specific instrument of health-related quality of life. It contains 59 items measuring 8 domains (i.e., strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion. memory and thinking and participation) with a single item assessing perceived overall recovery from stroke. Items are rated on a 5-point Likert scale with lower scores indicating greater difficulty in task completion during the past week. The reliability, validity, and responsiveness have been shown to be satisfactory in stroke patients.
Change scores of Revised Nottingham Sensory Assessment (rNSA) | Baseline, and 4 weeks
  The rNSA includes tactile sensation, kinesthetic sensation, and stereognosis. The rNSA is reliable measure of sensory function in stroke patients. For tactile sensation, the patient will be asked to indicate whenever he or she feels the test sensation. For kinesthetic sensations, all 3 aspects of movement will be tested: appreciation of movement, its direction and accurate joint position sense. The limb on the affected side of the body will be supported and moved by the examiner in various directions but movement is only at one joint at a time. The patients will be asked to mirror the change of movement with the other limb. For stereognosis, the object will be placed in the patient's hand for a maximum of 30 seconds. Identification is by naming, description or by pair-matching with an identical set. The object may be moved around the affected hand by the examiner. The rNSA has good intrarater and interrater reliability (Lincoln, Jackson, & Adams, 1998).

SECONDARY OUTCOMES:
Change scores of Adelaide Activities Profile (AAP) | Baseline, and 4 weeks, 16 weeks, and 28 weeks
  AAP will be applied to indicate the level of participation in household and community activities. This profile includes 21 activities in the four areas: domestic chores, household maintenance, service to others, and social activities. It scores on a scale of 0-3, with higher point meaning more frequent participation. The AAP is found to have good validity and reliability (Bond & Clark, 1998). The Nottingham Extended Activities of Daily Living (NEADL) Scale (Nouri, & Lincoln, 1987) is frequently used in clinical practice and research in rehabilitation to assess patients' independence in activities of daily living. Twenty-two activities are considered, which full in to 4 subscales: mobility, kitchen, domestic, and leisure activity. Responses are using 1 of 4 options (0 = not at all, 1 = with help, 2 = on my own with difficulty, 3 = on my own).
Change scores of 10-Meter Walk Test (10MWT) | Baseline, 4 weeks
  The 10MWT assess mobility function by measuring the time and the numbers of strides required to walk 10 meters under two conditions: (1) with the self-pace of each participant (self-pace); (2) with the speed that the participants walked as soon as possible. The velocity and stride length of the participant are calculated. Research has validated the 10MWT in measuring mobility in stroke.
Change scores of Actigraphy | Baseline, and 4 weeks
  The activity monitors will be used to provide a direct and objective measure of the amount of the impaired arm movement outside the laboratory. This measure, quantitatively recording the amount of activity in free-living conditions, will be used to reflect increase in the amount of affected arm use over time. The participants will be asked to wear an activity monitor, Actigraphy (Ambulatory Monitoring Inc., New York), on each wrist for 3 consecutive days to measure what amount they actually do in their daily life before and immediately after treatment. The Actigraphy can be attached to the subject's limb and measures the motion of that limb through an accelerometer. In this project, acceleration will be sampled at 10 Hz and summed over a user-specified epoch. The recording epoch will be 2 seconds; recording capacity will be approximately 72 hours. The ratio of affected to non-affected arm movement is a reliable and valid real-life measure of treatment outcome.
Change scores of Kinematic analysis | Baseline, and 4 weeks
  The kinematic analysis will involve unilateral and bilateral tasks, in which the participants will be asked to perform by using the affected upper limb or both upper limb simultaneously. A motion analysis system with 7 cameras (VICON MX 30d, Oxford Metrics Inc., Oxford, UK) will be used to capture the motion of arm (s) in kinematic testing. The markers will be attached on the styloid processes of the ulna. Depending on the unilateral or bilateral tasks, the makers will be placed on the affected arm or the both arms, respectively.
Change scores of hand strength | Baseline, 2 weeks, and 4 weeks
  The Baseline digital hydraulic hand dynamometer and pinch gauge (Fabrication Enterprises Inc, NY.) were used for measurement of grip and pinch strength. For the grip strength measurement, participants were instructed to squeeze the dynamometer with their hand as hard as they could. For the lateral pinch strength measurement, the pinch gauge was positioned between the pad of the thumb and the radial side of the middle phalanx of the index finger. For palmar pinch strength measurement, the pinch gauge was grasped between the pad of the thumb and the pad of the index finger. Participants were told to pinch as hard as they could. This method shows high repeatability (Haidar, Kumar, Bassi, & Deshmukh, 2004).
Change scores of Stroop test | Baseline, and 4 weeks
  The Number Stroop Test of the Psychology Experiment Building Language (Mueller, & Piper, 2014) was used to assess the inhibition ability. Participants will be asked to respond to the amount but not the name of stimuli.
Change scores of pressure pain threshold | Baseline, and 4 weeks
  The Commander Algometer (JTECH Medical, USA) is designed for easy handling and fine resolution to identify clinically significant pain sensitivity changes. The Commander Algometer provides a convenient, efficient, objective pain evaluation tool for treatment planning, progress evaluation and case management. The measured pressure thresholds/tolerances and trigger point tenderness will be reported by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (4):
- Taiwan (4):
  - Yong Cheng Rehabilitation Clinic, Taipei
  - Xing Cheng Rehabilitation Clinic, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
  - Lo-Sheng Sanatorium and Hospital, Taoyuan District

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411